CLINICAL TRIAL: NCT02746003
Title: Health Impacts of a Climate Change Adaptation Strategy to Address Drinking-water Salinity in Coastal Bangladesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Dhaka (Other); University College, London (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PR-15096
Record Dates: First submitted 2016-04-03; First posted 2016-04-21 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2017-09

CONDITIONS: Hypertension
Keywords: drinking water; salinity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Managed Aquifer Recharge water (Other): All the study population will receive the intervention by a random allocation over the study period. The study participants will be in both intervention and control at different times.
  Interventions: Other: Managed Aquifer Recharge water
- Control (Other): All the study population will receive the intervention by a random allocation over the study period. The study participants will be in both intervention and control arms at different times.
  Interventions: Other: Managed Aquifer Recharge water

INTERVENTIONS:
Other: Managed Aquifer Recharge water — Rain water will be recharged through slow sand filter and recharge wells into the confined underground aquifer and the surrounding community will abstract the water for drinking and cooking purposes

SUMMARY:
Background (brief):

1. Burden:

   Excessive salinity is common in groundwater aquifers across south-western coastal Bangladesh. Higher adult mean systolic and diastolic blood pressure and increased risk of gestational hypertension has been observed among those who drank tube-well water with high sodium content.
2. Knowledge gap:

   Managed Aquifer Recharge (MAR) systems, that inject freshwater into shallow aquifers, reduce drinking water salinity, have been successfully installed in the south-western area, providing year-round freshwater. However, the health benefits and risks of MAR water have not been measured.
3. Relevance:

If drinking MAR water can reduce hypertension in adults and pregnant women, while showing minimal risk of microbiological and chemical contamination, scale up can be considered.

Hypothesis (if any):

Mean systolic and diastolic blood pressure will be lower among the adult population who drink MAR water compared to people drinking saline or brackish groundwater Objectives: To determine

1. If providing access to MAR water for drinking and food preparation reduces blood pressure among the adult population > 20 years of age.
2. If providing access to MAR water for drinking and food preparation during pregnancy can reduce blood pressure among pregnant women.
3. If MAR water is contaminated with E coli and fecal coliforms.
4. Whether the MAR water is contaminated with dissolved constituents mobilized from aquifer sediments that are known to be harmful to human health.

Methods:

A stepped-wedge RCT will be conducted among communities before and after the intervention roll out. Study investigators will collect baseline information from all sites in the first monthly block (step) when no one will drink MAR water. There will be promoters who will convey messages regarding exclusive use of MAR water for drinking and cooking, at home and elsewhere. Measurements will be made by trained research assistants once every month. MAR water, pond water, groundwater and household stored water samples will be collected and tested once every month.

DETAILED DESCRIPTION:
Study sites:

The proposed study will be a stepped-wedge RCT that will be implemented in 20 MAR communities All 20 MAR communities will gradually have access to MAR water, but their access will be at different time periods or steps. Therefore, each MAR site will contribute data for both the intervention and the control time periods. There will be five, monthly steps in the stepped wedge trial. In the first monthly step, none of the communities will have MAR water available for drinking and the baseline information will be collected from all communities. During each subsequent month, five MAR communities will be randomly assigned to receive the intervention. In the last (fifth) monthly step, all the communities will have access to MAR drinking water. Blood pressure of all enrolled participants will be measured during each step. Animal and human studies suggest change in salt load changes blood pressure within few hours, and a meta-analysis of randomized trials suggest modest reduction in salt intake for four or more weeks causes significant reduction in blood pressure at the population-level. Therefore, the investigators will use an interval of at least one month between access to MAR water and first post-intervention blood pressure measurement, and between two consecutive blood pressure measurements.

This study protocol has been approved by the icddr,b Ethical Review Committee. Informed written consent will be taken from all participants and household heads.

Site selection and randomization:

The 30 MAR communities that are ready to roll out intervention (access to MAR water to the community) are located in rural areas in the three districts and 20 MAR communities which can be reached most effectively based on geographical location will be selected. Water samples from the selected 20 MAR sites will be collected every month for one year from June, 2016 to May, 2017 to capture the seasonal variation of microbiological and chemical water quality. Human health data and biological specimens from the enrolled participants from within the catchment area of the selected 20 sites will be collected from December, 2016 to May, 2017.

Sample Size Calculation The sample size of the stepped wedge trial was calculated based on the primary objective: reduction of systolic blood pressure. Data from southwest Bangladesh suggest a 7 mmHg lower mean systolic blood pressure among pregnant women who drank pond water compared to those who drank brackish water, and a 17 mmHg lower mean systolic blood pressure for pregnant women who drank rainwater compared to those who drank brackish water. The mean reduction in systolic blood pressure following long term modest salt reduction is 4.2 mmHg. At least three mmHg of systolic blood pressure reduction has been considered for the current study among the communities who will have access to MAR water for drinking and cooking purposes compared to those who will use brackish water. The entire population under the catchment area of an MAR community will be considered as one cluster. Each MAR community serves approximately 300 people, constituting 60-70 households in the catchment area. The mean household size in southwest coastal Bangladesh is 4.2; approximately 52% of household members are ≥ 20 years. Since blood pressure will be collected for all household members ≥ 20 years, an average of 2.2 participants has been estimated to be in this age group per household. About 28 households per cluster (28 *2.2 = 60 people per cluster) will be selected for the study. A previously published study in Bangladesh reported standard deviation (SD) for systolic blood pressure as 13.51. The sample size of the stepped wedge trial has been estimated adopting the formula used by Woertman et al. 2013 and Hemming et al. 2015. Woertman et al. proposed the usual approach of initially calculating the sample size for a simple unadjusted trial (NU), and then multiplying by the design effect for stepped wedge trial (DESW). The sample size of simple unadjusted trial was 1,868 participants (effect size= 3, standard deviation of 20 for both groups, 80% power, and 5% Type I error). The DESW was 3.046 based on formula provided by Woertman et al 2013. Considering a fixed cluster size of 60 and 5% loss-to-follow up, the proposed study will need 20 MAR communities, with five communities randomized to access MAR water in each step.

Sample size calculation for the pregnant women:

The mean SBP of the pregnant women south-western coastal Bangladesh is 102.4 mmHg among individuals who drank rainwater, 112.7 mmHg among filter users, 112.6 among pond water users and 119.4 among brackish groundwater users (tube-well water). The investigators assumed that drinking tube-well water may correspond with the dry season information and rainwater data correspond to the wet season information. Therefore, the assumption is that drinking MAR water would be able to reduce 17 mm Hg of systolic blood pressure. Considering crude birth rate of 26/1000 population, the assumption is there may be 88 birth during the seven months duration of the proposed study. Considering 88 pregnancies, the investigators will have 95% power to detect the effect of MAR in our main study. Stata command: sampsi 119.4 102.4, sd1(26.7) sd2(16.2) n1(44) n2(44) Data Analysis Blood Pressure The investigators will conduct an intention-to-treat analysis. Since the data will be longitudinal and on individual participants, generalized estimating equations (GEE) will be used with an appropriate autoregressive correlation structure, to account for repeated measures within individual study participants, and robust standard errors to allow for possible misspecification of the variance structure. The outcome is continuous blood pressure, which will be regressed on an indicator variable for access to MAR water, and dummy variables for the study sites to account for mean differences between communities... The interpretation of such a GEE model's output is the population average association of MAR with blood pressure, conditional on study site. The study investigators will further adjust for age, sex, body mass index, smoking, alcohol intake, family history of hypertension, and hypertensive medication of the participants. In secondary analyses, the association between drinking MAR water and urinary sodium and protein concentrations will be evaluated. For the pregnant women, we will control for the gestational week.

Water Quality Metrics T-test will be done to compare the microbial water quality as measured by the mean log10 MPN count/100 ml water during each monthly step between the MAR water and nearby pond water samples. The investigators will determine whether the concentration of each chemical constituent in water samples during each monthly step exceed the WHO recommended level. We will use similar GEE models as above for the outcomes of the log10 MPN count/100 ml water, and natural log-transformed (if skewed) concentration of each chemical constituent of water.

Referral of hypertensive patients- If research staff members identify hypertensive patients or cases of hypertensive disorders during pregnancy, they will refer patients to the government health facilities for further management. In addition, research staff will train pregnant women and family members to recognize the danger signs during pregnancy, and will also instruct them where to seek medical care if such danger signs appear. During household visits research staff will encourage pregnant women to attend prenatal visits.

Data management All data will be protected confidentially and only delinked personal information dataset will be used for analysis. The delinked dataset will be publicly available following publication of the primary result of the trial.

Collaborative Arrangements This project was co-developed by scientists affiliated with icddr,b, Emory University, Dhaka University, University College London, and Stanford University and has been funded by the Wellcome Trust, Our Planet, Our Health Award (GR 01336).. icddr,b will be responsible for implementing the protocol, collecting the data, and in collaboration with partner analyzing and reporting the results.

ELIGIBILITY:
Inclusion Criteria:

* Participants >20 years (both male and female)
* Pregnant women

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
reduction of mean systolic blood pressure among the >20 populations | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Md. Mahbubur Rahman, Principal Investigator — International Center for Diarrhoeal Disease Research, Bangladesh (icddr,b)
Locations (1):
- Dr. Md. Mahbubur Rahman, Dhaka, Bangladesh

REFERENCES:
- [Derived] Naser AM, Unicomb L, Doza S, Ahmed KM, Rahman M, Uddin MN, Quraishi SB, Selim S, Shamsudduha M, Burgess W, Chang HH, Gribble MO, Clasen TF, Luby SP. Stepped-wedge cluster-randomised controlled trial to assess the cardiovascular health effects of a managed aquifer recharge initiative to reduce drinking water salinity in southwest coastal Bangladesh: study design and rationale. BMJ Open. 2017 Sep 1;7(9):e015205. doi: 10.1136/bmjopen-2016-015205. PMID 28864689